CLINICAL TRIAL: NCT00896532
Title: A Randomised, Placebo-controlled, Multi-dose Phase 2 Study to Determine the Efficacy, Safety and Tolerability of AMG 785 in the Treatment of Postmenopausal Women With Low Bone Mineral Density
Brief Title: Romosozumab (AMG 785) in Postmenopausal Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060326; 2008-005991-28 (EudraCT Number)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Low Bone Mineral Density; Postmenopausal Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis, Postmenopausal | interventions — Alendronate; Teriparatide; romosozumab; Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo (Placebo Comparator): Participants received placebo matching to romosozumab once a month (QM) or once every 3 months (Q3M) administered subcutaneously (SC) for up to 24 months.
  Participants were then rerandomized to receive denosumab 60 mg or placebo to denosumab subcutaneously every 6 months from months 24 to 36. From months 36 to 48 participants received romosozumab 210 mg SC QM. At month 48 eligible participants received a single dose of open-label zoledronic acid 5 mg intravenously, or no intervention.
  Interventions: Drug: Placebo to Romosozumab; Drug: Denosumab; Drug: Placebo to Denosumab; Drug: Zoledronic acid
- Alendronate (Active Comparator): Participants received open-label alendronate (ALN) 70 mg orally (PO) every week (QW) for 12 months. At month 12 participants transitioned to receive romosozumab 140 mg subcutaneously every month for an additional 12 months (months 12 to 24).
  Participants were then rerandomized to receive denosumab 60 mg or placebo to denosumab subcutaneously every 6 months from months 24 to 36. At month 36 participants ended study participation.
  Interventions: Drug: Alendronate; Drug: Romosozumab; Drug: Denosumab; Drug: Placebo to Denosumab
- Teriparatide (Active Comparator): Participants received open-label teriparatide 20 μg subcutaneously every day (QD) for 12 months. At month 12 participants ended study participation.
  Interventions: Drug: Teriparatide
- Romosozumab 70 mg QM (Experimental): Participants received double-blind romosozumab 70 mg subcutaneously every month for 24 months.
  Participants were then rerandomized to receive denosumab 60 mg or placebo to denosumab subcutaneously every 6 months from months 24 to 36. From months 36 to 48 participants received romosozumab 210 mg SC QM. At month 48 eligible participants received a single dose of open-label zoledronic acid 5 mg intravenously, or no intervention.
  Interventions: Drug: Romosozumab; Drug: Denosumab; Drug: Placebo to Denosumab; Drug: Zoledronic acid
- Romosozumab 140 mg Q3M (Experimental): Participants received double-blind romosozumab 140 mg subcutaneously once every 3 months for 24 months.
  Participants were then rerandomized to receive denosumab 60 mg or placebo to denosumab subcutaneously every 6 months from months 24 to 36. From months 36 to 48 participants received romosozumab 210 mg SC QM. At month 48 eligible participants received a single dose of open-label zoledronic acid 5 mg intravenously, or no intervention.
  Interventions: Drug: Romosozumab; Drug: Denosumab; Drug: Placebo to Denosumab; Drug: Zoledronic acid
- Romosozumab 140 mg QM (Experimental): Participants received double-blind romosozumab 140 mg QM subcutaneously for 24 months.
  Participants were then rerandomized to receive denosumab 60 mg or placebo to denosumab subcutaneously every 6 months from months 24 to 36. From months 36 to 48 participants received romosozumab 210 mg SC QM. At month 48 eligible participants received a single dose of open-label zoledronic acid 5 mg intravenously, or no intervention.
  Interventions: Drug: Romosozumab; Drug: Denosumab; Drug: Placebo to Denosumab; Drug: Zoledronic acid
- Romosozumab 210 mg Q3M (Experimental): Participants received double-blind romosozumab 210 mg Q3M subcutaneously for 24 months.
  Participants were then rerandomized to receive denosumab 60 mg or placebo to denosumab subcutaneously every 6 months from months 24 to 36. From months 36 to 48 participants received romosozumab 210 mg SC QM. At month 48 eligible participants received a single dose of open-label zoledronic acid 5 mg intravenously, or no intervention.
  Interventions: Drug: Romosozumab; Drug: Denosumab; Drug: Placebo to Denosumab; Drug: Zoledronic acid
- Romosozumab 210 mg QM (Experimental): Participants received double-blind romosozumab 210 mg QM subcutaneously for 24 months.
  Participants were then rerandomized to receive denosumab 60 mg or placebo to denosumab subcutaneously every 6 months from months 24 to 36. From months 36 to 48 participants received romosozumab 210 mg SC QM. At month 48 eligible participants received a single dose of open-label zoledronic acid 5 mg intravenously, or no intervention.
  Interventions: Drug: Romosozumab; Drug: Denosumab; Drug: Placebo to Denosumab; Drug: Zoledronic acid

INTERVENTIONS:
Drug: Placebo to Romosozumab — Administered by subcutaneous injection QM or Q3M.
  Arms: Placebo
Drug: Alendronate — Administered orally once a week
  Other Names: Fosamax
  Arms: Alendronate
Drug: Teriparatide — Teriparatide 20 μg administered by subcutaneous injection once a day
  Other Names: Forsteo
  Arms: Teriparatide
Drug: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; EVENITY™
  Arms: Alendronate; Romosozumab 140 mg Q3M; Romosozumab 140 mg QM; Romosozumab 210 mg Q3M; Romosozumab 210 mg QM; Romosozumab 70 mg QM
Drug: Denosumab — Denosumab 60 mg administered by subcutaneous injection Q6M
  Other Names: Prolia®
  Arms: Alendronate; Placebo; Romosozumab 140 mg Q3M; Romosozumab 140 mg QM; Romosozumab 210 mg Q3M; Romosozumab 210 mg QM; Romosozumab 70 mg QM
Drug: Placebo to Denosumab — Administered by subcutaneous injection Q6M
  Arms: Alendronate; Placebo; Romosozumab 140 mg Q3M; Romosozumab 140 mg QM; Romosozumab 210 mg Q3M; Romosozumab 210 mg QM; Romosozumab 70 mg QM
Drug: Zoledronic acid — Zoledronic acid 5 mg administered intravenously
  Other Names: Aclasta
  Arms: Placebo; Romosozumab 140 mg Q3M; Romosozumab 140 mg QM; Romosozumab 210 mg Q3M; Romosozumab 210 mg QM; Romosozumab 70 mg QM

SUMMARY:
The primary objective was to determine the effect of treatment with romosozumab versus placebo at month 12 on the percent change from baseline in bone mineral density (BMD) at the lumbar spine in postmenopausal women with low bone density.

DETAILED DESCRIPTION:
This study included a 24-month treatment phase followed by rerandomization to a 12-month extension phase with denosumab or placebo, followed by a 12-month retreatment phase with romosozumab, followed by a 24-month follow-on phase with zoledronic acid or no intervention.

* 24-month Romosozumab Treatment Phase (months 1 to 24): Participants were randomized in a 1:1:1:1:1:1:1:1 ratio to receive 1 of 5 double-blind dosing regimens of romosozumab or placebo or open-label alendronate (ALN) or open-label teriparatide (TPTD) for the first 12 months of the study. At month 12, participants in the romosozumab and placebo groups continued their assigned treatment for an additional 12 months, participants in the TPTD group ended study participation, and participants in the ALN group transitioned to receive romosozumab 140 mg subcutaneously (SC) every month (QM) for an additional 12 months (months 12 to 24).
* 12-month Denosumab Extension Phase (months 24 to 36): At the end of the 24-month romosozumab treatment phase, eligible participants were randomized 1:1 within their original treatment group to receive either denosumab or placebo every 6 months (Q6M) for 12 months.
* 12-month Romosozumab Retreatment Phase (months 36 to 48): From months 36 to 48, participants initially randomized to romosozumab or placebo received romosozumab 210 mg SC QM. Participants who initially received ALN ended their participation at month 36 and were not retreated with romosozumab.
* 24-month Follow-on Phase (months 48 to 72): At month 48, participants received 1 dose of zoledronic acid 5 mg intravenously or no intervention for an additional 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women, aged ≥ 55 to ≤ 85
* Low BMD measured by dual energy X-ray absorptiometry (DXA) and assessed by the central imaging vendor (equivalent to T-scores between -2.0 and -3.5)

Exclusion Criteria:

* History of vertebral fracture, or fragility fracture of the wrist, humerus, hip or pelvis after age 50
* Untreated hyper- or hypothyroidism
* Current hyper- or hypoparathyroidism, hypo- or hypercalcemia
* Elevated transaminases
* Significantly impaired renal function
* Positive for: human immunodeficiency virus (HIV), hepatitis-C or hepatitis-B surface antigen
* Malignancy
* History of solid organ or bone marrow transplants
* Use of agents affecting bone metabolism
* Contraindicated or intolerant of alendronate therapy
* Contraindicated or intolerant of teriparatide therapy

Inclusion Criteria for the 12 month extension phase (Month 24 to 36):

- Normocalcemia at or after the Month 21 visit but before the Month 24 study visit

Exclusion Criteria for the 12 month extension phase (Month 24 to 36)

* Incidence of a clinical vertebral fracture or fragility fracture of the wrist, humerus, hip or pelvis during the initial 24 month treatment phase of the study
* A BMD loss of ≥ 7.0% from baseline at any time up to the Month 18 visit of the initial 24-month treatment phase
* Malignancy
* History of osteonecrosis of the jaw
* Use of proscribed medication during the initial 24 month treatment phase
* Contraindicated or intolerant of denosumab therapy

Inclusion Criteria for the 12 month re-treatment phase (Month 36 to 48)

* Albumin adjusted serum calcium of the most recent blood draw at or after the Month 30 visit but before the Month 36 study visit. Calcium repletion is permitted and central laboratory analysis of albumin adjusted serum calcium may be repeated before the Month 36 study visit
* Participation in Group A or B during initial 24 month treatment phase
* Subject has reached M36 of the study
* Appropriate written informed consent must be obtained

Exclusion Criteria for the 12 month re-treatment phase (Month 36 to 48)

* New malignancy
* Use of proscribed medication during the 12 month extension phase

Inclusion Criteria for the 24 month follow-on phase (Month 48 to 72) General inclusion criteria for participation

* Subject has reached month 48 of the study
* Appropriate written informed consent must be obtained Inclusion criteria for assignment to the no intervention group
* During the 24 month AMG 785 treatment phase, subject was assigned to any AMG 785 treatment group
* During the 12 month denosumab extension phase, subject was assigned to the denosumab treatment group Exclusion for the 24 month follow-on phase (Month 48 to 72)
* New malignancy
* Use of proscribed meds during the 12 month re-treatment phase
* Partial informed consent withdrawal and discontinuation of investigational product at any time up to month 48 visit
* Incidence of a clinical vertebral fracture or fragility fracture of the wrist, humerus, hip or pelvis during the initial 24 month treatment phase of the study
* BMD T-score of ≤ -2.5 at the lumbar spine, total hip, or femoral neck based on local read of the DXA scans at month 48
* Intolerance to zoledronic acid

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2009-06-03 (Actual); Primary Completion 2011-02-21 (Actual); Study Completion 2016-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Genant HK, Engelke K, Bolognese MA, Mautalen C, Brown JP, Recknor C, Goemaere S, Fuerst T, Yang YC, Grauer A, Libanati C. Effects of Romosozumab Compared With Teriparatide on Bone Density and Mass at the Spine and Hip in Postmenopausal Women With Low Bone Mass. J Bone Miner Res. 2017 Jan;32(1):181-187. doi: 10.1002/jbmr.2932. Epub 2016 Sep 20. PMID 27487526
- [Background] Keaveny TM, Crittenden DB, Bolognese MA, Genant HK, Engelke K, Oliveri B, Brown JP, Langdahl BL, Yan C, Grauer A, Libanati C. Greater Gains in Spine and Hip Strength for Romosozumab Compared With Teriparatide in Postmenopausal Women With Low Bone Mass. J Bone Miner Res. 2017 Sep;32(9):1956-1962. doi: 10.1002/jbmr.3176. Epub 2017 Jun 26. PMID 28543940
- [Background] Kendler DL, Bone HG, Massari F, Gielen E, Palacios S, Maddox J, Yan C, Yue S, Dinavahi RV, Libanati C, Grauer A. Bone mineral density gains with a second 12-month course of romosozumab therapy following placebo or denosumab. Osteoporos Int. 2019 Dec;30(12):2437-2448. doi: 10.1007/s00198-019-05146-9. Epub 2019 Oct 18. PMID 31628490
- [Background] McClung MR, Brown JP, Diez-Perez A, Resch H, Caminis J, Meisner P, Bolognese MA, Goemaere S, Bone HG, Zanchetta JR, Maddox J, Bray S, Grauer A. Effects of 24 Months of Treatment With Romosozumab Followed by 12 Months of Denosumab or Placebo in Postmenopausal Women With Low Bone Mineral Density: A Randomized, Double-Blind, Phase 2, Parallel Group Study. J Bone Miner Res. 2018 Aug;33(8):1397-1406. doi: 10.1002/jbmr.3452. Epub 2018 May 22. PMID 29694685
- [Background] McClung MR, Bolognese MA, Brown JP, Reginster JY, Langdahl BL, Maddox J, Shi Y, Rojeski M, Meisner PD, Grauer A. A single dose of zoledronate preserves bone mineral density for up to 2 years after a second course of romosozumab. Osteoporos Int. 2020 Nov;31(11):2231-2241. doi: 10.1007/s00198-020-05502-0. Epub 2020 Jul 4. PMID 32623487
- [Background] McClung MR, Bolognese MA, Brown JP, Reginster JY, Langdahl BL, Shi Y, Timoshanko J, Libanati C, Chines A, Oates MK. Skeletal responses to romosozumab after 12 months of denosumab. JBMR Plus. 2021 Jun 3;5(7):e10512. doi: 10.1002/jbm4.10512. eCollection 2021 Jul. PMID 34258507
- [Background] Poole KE, Treece GM, Pearson RA, Gee AH, Bolognese MA, Brown JP, Goemaere S, Grauer A, Hanley DA, Mautalen C, Recknor C, Yang YC, Rojeski M, Libanati C, Whitmarsh T. Romosozumab Enhances Vertebral Bone Structure in Women With Low Bone Density. J Bone Miner Res. 2022 Feb;37(2):256-264. doi: 10.1002/jbmr.4465. Epub 2021 Dec 16. PMID 34738660
- [Derived] McClung MR, Grauer A, Boonen S, Bolognese MA, Brown JP, Diez-Perez A, Langdahl BL, Reginster JY, Zanchetta JR, Wasserman SM, Katz L, Maddox J, Yang YC, Libanati C, Bone HG. Romosozumab in postmenopausal women with low bone mineral density. N Engl J Med. 2014 Jan 30;370(5):412-20. doi: 10.1056/NEJMoa1305224. Epub 2014 Jan 1. PMID 24382002
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 29 centers in 7 countries in Europe, North America, and Argentina. Participants were enrolled from the 3rd of June 2009 to the 17th of February 2010.
Pre-assignment Details: A total of 807 patients were screened and 419 were randomized. The study included a 24-month treatment phase, followed by rerandomization to a 12-month extension phase with denosumab or placebo; followed by a 12-month retreatment phase with romosozumab, followed by a 24-month follow-on phase with zoledronic acid or no intervention.
Groups:
- Placebo: Participants received placebo matching to romosozumab once a month (QM) or once every 3 months (Q3M) administered subcutaneously for 24 months.
- Alendronate: Participants received open-label alendronate (ALN) 70 mg orally (PO) every week (QW) for 12 months. At month 12 participants transitioned to receive romosozumab 140 mg subcutaneously every month for an additional 12 months (months 12 to 24).
- Romosozumab 70 mg QM: Participants received double-blind romosozumab 70 mg subcutaneously every month for 24 months.
- Romosozumab 140 mg Q3M: Participants received double-blind romosozumab 140 mg subcutaneously once every 3 months for 24 months.
- Romosozumab 140 mg QM: Participants received double-blind romosozumab 140 mg QM subcutaneously for 24 months.
- Romosozumab 210 mg Q3M: Participants received double-blind romosozumab 210 mg Q3M subcutaneously for 24 months.
- Romosozumab 210 mg QM: Participants received double-blind romosozumab 210 mg QM subcutaneously for 24 months.
- Month 24-36: Placebo/Placebo: Participants who received placebo in the 24-month romosozumab treatment phase then received placebo to denosumab subcutaneously once every 6 months (Q6M) for 12 months during the denosumab extension phase.
- Month 24-36: Placebo/Denosumab: Participants who received placebo in the 24-month romosozumab treatment phase then received denosumab 60 mg subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 24-36: Alendronate/Romosozumab/Placebo: Participants who received alendronate for the first 12 months and romosozumab 140 mg subcutaneously every month from months 12 to 24 received placebo to denosumab subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 24-36: Alendronate/Romosozumab/Denosumab: Participants who received alendronate for the first 12 months, romosozumab 140 mg subcutaneously QM from months 12 to 24 received denosumab 60 mg subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 24-36: Romosozumab/Placebo: Participants who received romosozumab at any dose for 24 months in the romosozumab treatment phase received placebo to denosumab subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 24-36: Romosozumab/Denosumab: Participants who received romosozumab at any dose for 24 months in the romosozumab treatment phase received denosumab 60 mg subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 36-48: Placebo/Placebo/Romosozumab: Participants who received placebo in the first 24-month romosozumab treatment phase and placebo to denosumab during months 24-36 then received romosozumab 210 mg subcutaneously QM in the 12-month romosozumab retreatment phase (months 36 to 48).
- Month 36-48: Placebo/Denosumab/Romosozumab: Participants who received placebo in the first 24 month romosozumab treatment phase and denosumab 60 mg during months 24 to 36 then received romosozumab 210 mg subcutaneously QM in the 12-month romosozumab retreatment phase (months 36 to 48).
- Month 36-48: Romosozumab/Placebo/Romosozumab: Participants who received romosozumab at any dose during the first 24-month romosozumab treatment phase and placebo to denosumab during months 24 to 36 then received romosozumab 210 mg subcutaneously QM in the 12-month romosozumab retreatment phase (months 36 to 48).
- Month 36-48: Romosozumab/Denosumab/Romosozumab: Participants who received romosozumab at any dose during the first 24-month romosozumab treatment phase and denosumab 60 mg during months 24 to 36 then received romosozumab 210 mg subcutaneously QM in the 12-month romosozumab retreatment phase (months 36 to 48).
- Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention: Participants who received romosozumab at any dose during the 24-month romosozumab treatment phase, denosumab 60 mg during months 24 to 36 and romosozumab 210 mg QM in months 36 to 48 then received no intervention during the 24-month follow-on phase (months 48-72).
- Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid: Participants who received placebo in the 24-month romosozumab treatment phase, placebo to denosumab during months 24 to 36 and romosozumab 210 mg QM in months 36 to 48 then received a single dose of open-label zoledronic acid 5 mg intravenously at month 48.
- Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic Acid: Participants who received placebo in the 24-month romosozumab treatment phase, denosumab 60 mg Q6M from months 24 to 36 and romosozumab 210 mg QM from months 36 to 48 then received a single dose of open-label zoledronic acid 5 mg intravenously at month 48.
- Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid: Participants who received romosozumab at any dose during the 24-month romosozumab treatment phase, placebo to denosumab during months 24 to 36 and romosozumab 210 mg QM in months 36 to 48 then received a single dose of open-label zoledronic acid 5 mg intravenously at month 48.
- Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid: Participants who received romosozumab at any dose during the 24-month romosozumab treatment phase, denosumab 60 mg Q6M during months 24 to 36 and romosozumab 210 mg QM in months 36 to 48 then received a single dose of open-label zoledronic acid 5 mg intravenously at month 48.
Period: Months 1-24: Romosozumab Treatment Phase
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM | Month 24-36: Placebo/Placebo | Month 24-36: Placebo/Denosumab | Month 24-36: Alendronate/Romosozumab/Placebo | Month 24-36: Alendronate/Romosozumab/Denosumab | Month 24-36: Romosozumab/Placebo | Month 24-36: Romosozumab/Denosumab | Month 36-48: Placebo/Placebo/Romosozumab | Month 36-48: Placebo/Denosumab/Romosozumab | Month 36-48: Romosozumab/Placebo/Romosozumab | Month 36-48: Romosozumab/Denosumab/Romosozumab | Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention | Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid
Started | 52 | 51 | 55 | 51 | 54 | 51 | 53 | 52 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 51 (One participant received 1 dose of romosozumab 70 mg in error) | 51 | 54 | 49 | 53 | 48 | 53 | 51 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed 12 Months | 47 | 49 | 46 | 45 | 50 | 46 | 51 | 49 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 46 | 45 | 46 | 39 | 46 | 43 | 48 | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 9 | 12 | 8 | 8 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 4 | 6 | 5 | 6 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — On-study But No Month 24 Visit | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Months 24-36: Denosumab Extension Phase
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM | Month 24-36: Placebo/Placebo | Month 24-36: Placebo/Denosumab | Month 24-36: Alendronate/Romosozumab/Placebo | Month 24-36: Alendronate/Romosozumab/Denosumab | Month 24-36: Romosozumab/Placebo | Month 24-36: Romosozumab/Denosumab | Month 36-48: Placebo/Placebo/Romosozumab | Month 36-48: Placebo/Denosumab/Romosozumab | Month 36-48: Romosozumab/Placebo/Romosozumab | Month 36-48: Romosozumab/Denosumab/Romosozumab | Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention | Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 20 | 21 | 93 | 90 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 (Includes one participant who received 1 dose of romosozumab 70 mg in error in first 12 months) | 19 | 19 | 90 | 88 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 18 | 18 | 19 | 88 | 88 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Months 36-48: Romosozumab Retreatment
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM | Month 24-36: Placebo/Placebo | Month 24-36: Placebo/Denosumab | Month 24-36: Alendronate/Romosozumab/Placebo | Month 24-36: Alendronate/Romosozumab/Denosumab | Month 24-36: Romosozumab/Placebo | Month 24-36: Romosozumab/Denosumab | Month 36-48: Placebo/Placebo/Romosozumab | Month 36-48: Placebo/Denosumab/Romosozumab | Month 36-48: Romosozumab/Placebo/Romosozumab | Month 36-48: Romosozumab/Denosumab/Romosozumab | Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention | Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 16 | 72 | 67 | 0 | 0 | 0 | 0 | 0
Received Romosozumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 16 (Includes one participant who received 1 dose of romosozumab 70 mg in error in first 12 months) | 72 | 67 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 14 | 65 | 64 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Continuing the re-treatment phase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Months 48-72: Follow-on Phase
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM | Month 24-36: Placebo/Placebo | Month 24-36: Placebo/Denosumab | Month 24-36: Alendronate/Romosozumab/Placebo | Month 24-36: Alendronate/Romosozumab/Denosumab | Month 24-36: Romosozumab/Placebo | Month 24-36: Romosozumab/Denosumab | Month 36-48: Placebo/Placebo/Romosozumab | Month 36-48: Placebo/Denosumab/Romosozumab | Month 36-48: Romosozumab/Placebo/Romosozumab | Month 36-48: Romosozumab/Denosumab/Romosozumab | Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention | Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 51 | 11 | 12 | 59 | 8
Received Zoledronic Acid | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 12 | 56 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 11 | 12 | 57 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Ineligibility Determined | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants (full analysis set)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM | Total
Number analyzed (Participants) | 52 | 51 | 55 | 51 | 54 | 51 | 53 | 52 | 419
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (6.5) | 67.1 (5.8) | 66.8 (5.7) | 65.8 (6.1) | 67.3 (6.7) | 67.8 (6.2) | 66.1 (7.3) | 66.3 (6.5) | 66.8 (6.4)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 20 | 18 | 21 | 21 | 20 | 12 | 24 | 18 | 154
  ≥ 65 years | 32 | 33 | 34 | 30 | 34 | 39 | 29 | 34 | 265
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 55 | 51 | 54 | 51 | 53 | 52 | 419
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 47 | 46 | 44 | 46 | 43 | 48 | 44 | 44 | 362
  Black or African American | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
  Hispanic or Latino | 5 | 4 | 9 | 5 | 8 | 3 | 8 | 6 | 48
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 4
  Japanese | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lumbar Spine Bone Mineral Density (BMD) T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. A normal T-score is -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.29 (0.66) | -2.08 (0.69) | -2.29 (0.57) | -2.35 (0.79) | -2.44 (0.70) | -2.27 (0.77) | -2.21 (0.69) | -2.33 (0.57) | -2.29 (0.68)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] | -1.35 (0.67) | -1.55 (0.68) | -1.32 (0.78) | -1.69 (0.67) | -1.58 (0.51) | -1.67 (0.65) | -1.65 (0.63) | -1.45 (0.65) | -1.53 (0.66)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: T-score] | -1.76 (0.56) | -1.91 (0.61) | -1.79 (0.67) | -2.06 (0.55) | -2.00 (0.54) | -2.03 (0.58) | -2.02 (0.57) | -1.87 (0.58) | -1.93 (0.59)
Distal 1/3 Radius BMD T-score [Mean (Standard Deviation); unit: T-score] — Population: Participants with available data
  T-score
    number analyzed (Participants) | 51 | 50 | 50 | 49 | 52 | 47 | 52 | 49 | 400
    (all) | -1.85 (1.04) | -2.08 (0.99) | -2.05 (1.21) | -1.78 (1.14) | -2.24 (1.06) | -2.11 (1.12) | -1.98 (1.04) | -2.03 (0.99) | -2.01 (1.08)
Serum Type 1 Collagen C-telopeptide (CTX) [Median (Inter-Quartile Range); unit: ng/L] — Population: Participants with available data
  ng/L
    number analyzed (Participants) | 51 | 51 | 54 | 49 | 53 | 48 | 53 | 51 | 410
    (all) | 481.0 [347.0 to 673.0] | 494.0 [373.0 to 614.0] | 505.5 [410.0 to 690.0] | 486.0 [374.0 to 627.0] | 525.0 [358.0 to 714.0] | 532.0 [363.0 to 621.5] | 478.0 [362.0 to 695.0] | 519.0 [405.0 to 642.0] | 501.5 [379.0 to 649.0]
Serum Procollagen Type 1 N-telopeptide (P1NP) [Median (Inter-Quartile Range); unit: μg/L] — Population: Participants with available data
  μg/L
    number analyzed (Participants) | 51 | 51 | 54 | 49 | 53 | 48 | 53 | 51 | 410
    (all) | 47.76 [37.92 to 59.12] | 49.25 [40.05 to 57.73] | 48.78 [42.45 to 66.98] | 50.36 [36.43 to 61.39] | 48.63 [37.55 to 67.47] | 48.13 [38.45 to 56.30] | 49.24 [39.57 to 62.16] | 52.58 [42.47 to 63.91] | 49.37 [39.57 to 61.86]
Osteocalcin [Median (Inter-Quartile Range); unit: ng/mL] — Population: Participants with available data
  ng/mL
    number analyzed (Participants) | 51 | 51 | 54 | 49 | 53 | 48 | 53 | 51 | 410
    (all) | 17.95 [15.78 to 23.62] | 19.37 [14.69 to 24.78] | 19.47 [15.93 to 26.14] | 19.03 [15.10 to 23.63] | 19.93 [14.92 to 26.72] | 18.56 [15.20 to 21.92] | 17.72 [13.61 to 23.16] | 18.36 [16.15 to 28.32] | 18.84 [15.13 to 24.16]
Bone-specific Alkaline Phosphatase (BSAP) [Median (Inter-Quartile Range); unit: μg/L] — Population: Participants with available data
  μg/L
    number analyzed (Participants) | 51 | 51 | 54 | 49 | 53 | 48 | 53 | 51 | 410
    (all) | 11.79 [9.75 to 13.53] | 12.93 [10.48 to 15.52] | 13.34 [10.04 to 16.39] | 11.82 [10.66 to 15.34] | 13.19 [10.10 to 15.68] | 11.78 [9.44 to 14.60] | 12.61 [10.06 to 14.04] | 12.37 [10.16 to 15.90] | 12.44 [10.06 to 15.30]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline at Month 12 in BMD at the Lumbar Spine
Description: Bone mineral density was measured using dual energy x-ray absorptiometry (DXA). Images were analyzed by a central imaging reader.
Time Frame: Baseline to 12 months
Population: All randomized participants who had non-missing baseline and month 12 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Romosozumab Monthly: Participants who received once a month dosing of romosozumab (70, 140 or 210 mg).
- Romosozumab Every 3 Months: Participants who received romosozumab every 3 months (140 or 210 mg)
- Romosozumab 140 mg: Participants who received romosozumab 140 mg dosing (QM or Q3M).
- Romosozumab 210 mg: Participants who received romosozumab 210 mg dosing (QM or Q3M).
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM | Romosozumab Monthly | Romosozumab Every 3 Months | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 47 | 47 | 46 | 44 | 49 | 46 | 51 | 49 | 139 | 100 | 95 | 100
percent change | -0.1 [-1.2 to 0.9] | 4.1 [3.0 to 5.1] | 7.1 [6.1 to 8.2] | 5.4 [4.3 to 6.4] | 5.4 [4.4 to 6.5] | 9.1 [8.0 to 10.2] | 5.5 [4.4 to 6.6] | 11.3 [10.3 to 12.4] | 8.6 [7.9 to 9.3] | 5.5 [4.7 to 6.3] | 7.3 [6.4 to 8.1] | 8.4 [7.6 to 9.2]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab Monthly; A linear mixed effects model was fit with the percent change from baseline to months 3, 6 and 12 in BMD of the lumbar spine as the dependent variable and baseline BMD, machine type, interaction of baseline BMD and machine type, geographic region (Latin America, North America, Europe), visit, treatment regimen (categorical), interaction of treatment regimen and visit as the independent variables; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model — P-value is adjusted by the Hochberg procedure for comparisons to placebo; LS Mean Difference from Placebo = 8.7, 95% CI 2-sided [7.5 to 9.9]
Statistical Analysis 2: Comparison: Placebo vs Romosozumab Every 3 Months; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model — P-value is adjusted by the Hochberg procedure for comparisons to placebo; LS Mean Difference from placebo = 5.6, 95% CI 2-sided [4.3 to 6.9]
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 140 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model — P-value is adjusted by the Hochberg procedure for comparisons to placebo; LS Mean Difference from Placebo = 7.4, 95% CI 2-sided [6.1 to 8.7]
Statistical Analysis 4: Comparison: Placebo vs Romosozumab 210 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model — P-value is adjusted by the Hochberg procedure for comparisons to placebo; LS Mean Difference from Placebo = 8.5, 95% CI 2-sided [7.3 to 9.8]

2. Secondary Outcome: Percent Change From Baseline at Month 6 in BMD at the Lumbar Spine
Description: Bone mineral density was measured using dual energy x-ray absorptiometry (DXA). Images were analyzed by a central imaging reader.
  Percent change from baseline to month 6 was analyzed using a linear mixed effects model with the percent change from baseline to month 6 in DXA BMD as dependent variable, and baseline BMD value, machine type, geographic region, interaction of baseline BMD and machine type, visit, treatment (categorical) and interaction of treatment and visit as the independent variables.
Time Frame: Baseline to 6 months
Population: All randomized participants who had non-missing baseline and month 6 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 49 | 49 | 48 | 43 | 49 | 47 | 52 | 50
percent change | 0.3 [-0.7 to 1.3] | 2.6 [1.6 to 3.6] | 4.8 [3.8 to 5.8] | 4.1 [3.1 to 5.1] | 4.2 [3.2 to 5.2] | 7.1 [6.1 to 8.1] | 4.4 [3.4 to 5.3] | 8.2 [7.3 to 9.2]

3. Secondary Outcome: Percent Change From Baseline at Month 6 in BMD of the Total Hip
Description: as for outcome 2
Time Frame: Baseline to 6 months
Population: All randomized participants who had non-missing baseline and month 6 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 49 | 49 | 48 | 43 | 49 | 47 | 52 | 50
percent change | -0.6 [-1.2 to -0.1] | 0.9 [0.3 to 1.5] | 0.5 [-0.0 to 1.1] | 0.5 [-0.1 to 1.1] | 0.9 [0.3 to 1.5] | 2.2 [1.7 to 2.8] | 1.1 [0.6 to 1.7] | 2.9 [2.3 to 3.4]

4. Secondary Outcome: Percent Change From Baseline at Month 6 in BMD of the Femoral Neck
Description: as for outcome 2
Time Frame: Baseline to 6 months
Population: All randomized participants who had non-missing baseline and month 6 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 49 | 49 | 48 | 43 | 49 | 47 | 52 | 50
percent change | -0.4 [-1.3 to 0.4] | 0.5 [-0.3 to 1.4] | 0.5 [-0.3 to 1.3] | 0.2 [-0.7 to 1.1] | 0.4 [-0.4 to 1.3] | 2.1 [1.3 to 3.0] | 0.9 [0.1 to 1.7] | 1.9 [1.0 to 2.7]

5. Secondary Outcome: Percent Change From Baseline at Month 12 in BMD of the Total Hip
Description: Bone mineral density was measured using dual energy x-ray absorptiometry (DXA). Images were analyzed by a central imaging reader.
  Percent change from baseline to 12 months in BMD was analyzed using a linear mixed effects model with the percent change from baseline to month 12 in DXA BMD as dependent variable, and baseline BMD value, machine type, geographic region, interaction of baseline BMD and machine type, visit, treatment (categorical) and interaction of treatment and visit as the independent variables.
Time Frame: Baseline to 12 months
Population: All randomized participants who had non-missing baseline and month 12 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 47 | 47 | 46 | 44 | 49 | 46 | 50 | 49
percent change | -0.7 [-1.4 to -0.1] | 1.9 [1.3 to 2.6] | 1.3 [0.7 to 2.0] | 1.3 [0.6 to 2.0] | 1.3 [0.7 to 2.0] | 3.4 [2.7 to 4.1] | 1.9 [1.3 to 2.6] | 4.1 [3.5 to 4.8]

6. Secondary Outcome: Percent Change From Baseline at Month 12 in BMD of the Femoral Neck
Description: as for outcome 5
Time Frame: Baseline to 12 months
Population: All randomized participants who had non-missing baseline and month 12 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 47 | 47 | 46 | 44 | 49 | 46 | 50 | 49
percent change | -1.1 [-2.0 to -0.2] | 1.2 [0.3 to 2.1] | 1.1 [0.2 to 2.0] | 0.6 [-0.3 to 1.6] | 1.8 [0.9 to 2.7] | 4.2 [3.3 to 5.1] | 1.4 [0.5 to 2.3] | 3.7 [2.8 to 4.6]

7. Secondary Outcome: Percent Change From Baseline at Month 12 in BMD of the Distal Radius
Description: Bone mineral density was measured using dual energy x-ray absorptiometry (DXA). Images were analyzed by a central imaging reader.
  Percent change from baseline in distal radius BMD was analyzed using an analysis of covariance (ANCOVA) model with the percent change from baseline to Month 12 in DXA BMD as dependent variable, baseline BMD value, machine type, interaction of baseline BMD and machine type, treatment (categorical) and geographic region as the independent class variables.
Time Frame: Baseline to 12 months
Population: All randomized participants who had non-missing baseline and month 12 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 48 | 46 | 42 | 44 | 48 | 46 | 49 | 46
percent change | -0.9 [-1.8 to 0.1] | -0.3 [-1.2 to 0.7] | -1.7 [-2.7 to -0.7] | -1.8 [-2.8 to -0.8] | -1.1 [-2.1 to -0.2] | -1.0 [-2.0 to -0.0] | -0.4 [-1.3 to 0.5] | -1.2 [-2.1 to -0.2]

8. Secondary Outcome: Percent Change From Baseline in Procollagen Type 1 N-telopeptide (P1NP)
Description: Percent change from baseline in the bone turnover marker (BTM) P1NP was analyzed using a linear mixed effects model with the natural logarithm of the ratio of BTM (follow-up versus baseline) as the dependent variables, and visit, treatment (categorical), interaction of treatment and visit and the natural logarithm of the baseline BTM as the independent variables; outcomes were then transformed back to percent change from baseline.
Time Frame: Baseline and months 1, 3, 6, 9, and 12
Population: All randomized participants with baseline and at least one post baseline measurement on or prior to the month 12 visit and with available data at each time point. Data were not collected for participants in the alendronate and teriparatide groups at month 1.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 50 | 51 | 49 | 49 | 53 | 48 | 53 | 50
percent change
  Month 1: number analyzed (Participants) | 50 | 0 | 0 | 49 | 52 | 48 | 52 | 50
  Month 1 | -0.7 [-8.7 to 8.1] |  |  | 24.2 [14.1 to 35.3] | 61.4 [48.6 to 75.3] | 55.0 [42.2 to 69.0] | 75.8 [61.8 to 90.9] | 92.2 [76.6 to 109.1]
  Month 3: number analyzed (Participants) | 50 | 51 | 49 | 48 | 52 | 48 | 52 | 50
  Month 3 | -5.4 [-13.6 to 3.6] | -50.8 [-55.1 to -46.2] | 97.1 [79.7 to 116.1] | -9.1 [-17.1 to -0.2] | -15.5 [-22.7 to -7.7] | 3.8 [-5.4 to 13.9] | -19.5 [-26.4 to -12.1] | 25.6 [14.6 to 37.5]
  Month 6: number analyzed (Participants) | 49 | 49 | 48 | 43 | 49 | 47 | 52 | 50
  Month 6 | -5.9 [-14.6 to 3.6] | -57.0 [-61.0 to -52.7] | 138.0 [115.7 to 162.6] | -20.0 [-27.7 to -11.4] | -22.8 [-29.9 to -15.0] | -18.6 [-26.3 to -10.1] | -25.5 [-32.2 to -18.1] | 6.9 [-3.0 to 17.8]
  Month 9: number analyzed (Participants) | 46 | 48 | 48 | 44 | 47 | 46 | 52 | 49
  Month 9 | -10.6 [-19.6 to -0.7] | -60.8 [-64.7 to -56.5] | 116.8 [95.1 to 140.9] | -26.9 [-34.4 to -18.5] | -23.8 [-31.4 to -15.4] | -26.1 [-33.6 to -17.8] | -30.1 [-36.8 to -22.6] | -5.8 [-15.1 to 4.6]
  Month 12: number analyzed (Participants) | 45 | 47 | 46 | 42 | 48 | 45 | 45 | 48
  Month 12 | -8.7 [-17.9 to 1.5] | -60.8 [-64.7 to -56.4] | 98.3 [78.3 to 120.5] | -23.0 [-31.0 to -14.0] | -23.3 [-30.9 to -14.9] | -31.2 [-38.2 to -23.4] | -29.7 [-36.7 to -22.1] | -17.2 [-25.4 to -8.1]

9. Secondary Outcome: Percent Change From Baseline in Type 1 Collagen C-telopeptide (CTX)
Description: Percent change from baseline in the bone turnover marker (BTM) CTX was analyzed using a linear mixed effects model with the natural logarithm of the ratio of BTM (follow-up versus baseline) as the dependent variables, and visit, treatment (categorical), interaction of treatment and visit and the natural logarithm of the baseline BTM as the independent variables; outcomes were then transformed back to percent change from baseline.
Time Frame: Baseline and months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 50 | 51 | 49 | 49 | 53 | 48 | 53 | 50
percent change
  Month 1: number analyzed (Participants) | 50 | 0 | 0 | 49 | 51 | 48 | 52 | 50
  Month 1 | -3.9 [-12.1 to 5.1] |  |  | -22.1 [-28.9 to -14.7] | -19.2 [-26.0 to -11.7] | -35.4 [-41.0 to -29.2] | -33.0 [-38.6 to -26.8] | -28.5 [-34.7 to -21.8]
  Month 3: number analyzed (Participants) | 50 | 46 | 49 | 48 | 52 | 48 | 52 | 50
  Month 3 | -2.4 [-12.0 to 8.2] | -65.0 [-68.5 to -61.1] | 69.4 [52.6 to 88.0] | -21.5 [-29.3 to -12.8] | -6.2 [-15.2 to 3.8] | -26.5 [-33.8 to -18.3] | -12.6 [-21.0 to -3.4] | -3.7 [-13.2 to 6.7]
  Month 6: number analyzed (Participants) | 49 | 47 | 48 | 43 | 48 | 46 | 52 | 50
  Month 6 | 2.7 [-8.4 to 15.2] | -64.2 [-68.1 to -59.8] | 93.5 [72.3 to 117.4] | -18.1 [-27.3 to -7.7] | -8.4 [-18.3 to 2.7] | -24.6 [-33.0 to -15.2] | -10.5 [-20.0 to 0.0] | -8.7 [-18.6 to 2.4]
  Month 9: number analyzed (Participants) | 46 | 47 | 48 | 43 | 47 | 46 | 52 | 49
  Month 9 | 1.0 [-11.2 to 14.9] | -64.4 [-68.6 to -59.5] | 81.3 [59.4 to 106.2] | -15.1 [-25.7 to -3.0] | 1.3 [-10.8 to 15.1] | -27.7 [-36.6 to -17.6] | -11.7 [-22.0 to -0.1] | -17.2 [-27.1 to -6.0]
  Month 12: number analyzed (Participants) | 45 | 45 | 46 | 42 | 48 | 45 | 45 | 48
  Month 12 | 9.8 [-3.9 to 25.4] | -66.7 [-70.8 to -62.0] | 77.0 [54.9 to 102.1] | -20.3 [-30.6 to -8.6] | 12.2 [-1.5 to 27.8] | -33.0 [-41.4 to -23.3] | -6.6 [-18.0 to 6.5] | -22.5 [-32.0 to -11.7]

10. Secondary Outcome: Percent Change From Baseline in Osteocalcin
Description: Percent change from baseline in the bone turnover marker (BTM) osteocalcin was analyzed using a linear mixed effects model with the natural logarithm of the ratio of BTM (follow-up versus baseline) as the dependent variables, and visit, treatment (categorical), interaction of treatment and visit and the natural logarithm of the baseline BTM as the independent variables; outcomes were then transformed back to percent change from baseline.
Time Frame: Baseline and months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 50 | 51 | 49 | 49 | 53 | 48 | 53 | 50
percent change
  Month 1: number analyzed (Participants) | 50 | 0 | 0 | 49 | 52 | 48 | 52 | 50
  Month 1 | -1.6 [-9.1 to 6.5] |  |  | 28.1 [18.3 to 38.7] | 60.1 [48.2 to 73.0] | 53.1 [41.2 to 65.9] | 77.9 [64.7 to 92.2] | 78.6 [65.0 to 93.2]
  Month 3: number analyzed (Participants) | 50 | 51 | 49 | 48 | 52 | 48 | 52 | 50
  Month 3 | 4.1 [-5.6 to 14.7] | -28.7 [-35.3 to -21.5] | 104.7 [85.5 to 125.9] | -0.3 [-9.8 to 10.1] | -5.6 [-14.2 to 3.8] | 15.6 [4.7 to 27.7] | -3.7 [-12.5 to 5.9] | 41.6 [28.4 to 56.1]
  Month 6: number analyzed (Participants) | 48 | 49 | 48 | 43 | 49 | 47 | 52 | 49
  Month 6 | -7.1 [-16.2 to 2.8] | -40.6 [-46.3 to -34.2] | 106.7 [86.5 to 129.1] | -11.8 [-20.8 to -1.8] | -16.5 [-24.5 to -7.6] | -7.4 [-16.5 to 2.8] | -23.2 [-30.5 to -15.3] | 10.0 [-0.7 to 21.7]
  Month 9: number analyzed (Participants) | 46 | 48 | 48 | 44 | 47 | 46 | 52 | 49
  Month 9 | -6.0 [-15.0 to 4.0] | -50.9 [-55.6 to -45.8] | 99.9 [80.8 to 121.0] | -26.9 [-34.1 to -18.9] | -29.0 [-35.8 to -21.6] | -27.7 [-34.7 to -19.9] | -30.7 [-37.1 to -23.7] | -4.0 [-13.1 to 6.0]
  Month 12: number analyzed (Participants) | 45 | 47 | 46 | 42 | 48 | 45 | 45 | 48
  Month 12 | -14.1 [-22.0 to -5.4] | -50.3 [-54.8 to -45.4] | 91.6 [74.1 to 110.9] | -27.3 [-34.1 to -19.6] | -24.7 [-31.4 to -17.2] | -31.1 [-37.5 to -24.1] | -26.2 [-32.9 to -18.9] | -12.5 [-20.4 to -3.9]

11. Secondary Outcome: Percent Change From Baseline in Bone-specific Alkaline Phosphatase (BSAP)
Description: Percent change from baseline in the bone turnover marker (BTM) BSAP was analyzed using a linear mixed effects model with the natural logarithm of the ratio of BTM (follow-up versus baseline) as the dependent variables, and visit, treatment (categorical), interaction of treatment and visit and the natural logarithm of the baseline BTM as the independent variables; outcomes were then transformed back to percent change from baseline.
Time Frame: Baseline and months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Alendronate | Teriparatide | Romosozumab 70 mg QM | Romosozumab 140 mg Q3M | Romosozumab 140 mg QM | Romosozumab 210 mg Q3M | Romosozumab 210 mg QM
Number analyzed (Participants) | 50 | 51 | 49 | 49 | 53 | 48 | 53 | 50
percent change
  Month 1: number analyzed (Participants) | 50 | 0 | 0 | 49 | 52 | 48 | 52 | 50
  Month 1 | -1.1 [-6.7 to 4.9] |  |  | 11.7 [5.2 to 18.5] | 35.1 [27.5 to 43.1] | 29.3 [21.8 to 37.3] | 47.5 [39.3 to 56.2] | 60.9 [51.7 to 70.7]
  Month 3: number analyzed (Participants) | 50 | 51 | 49 | 48 | 52 | 48 | 52 | 50
  Month 3 | -7.6 [-14.3 to -0.3] | -30.5 [-35.5 to -25.0] | 21.8 [12.8 to 31.4] | -8.5 [-15.3 to -1.1] | -18.0 [-23.9 to -11.7] | 1.3 [-6.2 to 9.4] | -17.3 [-23.2 to -10.9] | 27.4 [18.1 to 37.4]
  Month 6: number analyzed (Participants) | 48 | 49 | 48 | 43 | 49 | 46 | 52 | 49
  Month 6 | -4.1 [-12.1 to 4.5] | -35.4 [-40.8 to -29.7] | 29.8 [19.0 to 41.6] | -8.7 [-16.6 to -0.1] | -18.2 [-25.0 to -10.9] | -6.6 [-14.5 to 2.0] | -20.0 [-26.4 to -13.0] | 13.1 [3.8 to 23.3]
  Month 9: number analyzed (Participants) | 46 | 48 | 48 | 44 | 47 | 46 | 52 | 49
  Month 9 | 3.5 [-3.8 to 11.4] | -32.5 [-37.3 to -27.4] | 41.8 [31.7 to 52.6] | -4.9 [-11.9 to 2.6] | -12.5 [-18.7 to -5.9] | -5.5 [-12.3 to 1.8] | -17.7 [-23.3 to -11.7] | 10.4 [2.7 to 18.8]
  Month 12: number analyzed (Participants) | 45 | 47 | 46 | 42 | 48 | 45 | 45 | 48
  Month 12 | 9.2 [1.7 to 17.2] | -31.2 [-35.9 to -26.2] | 45.7 [35.7 to 56.4] | -2.6 [-9.5 to 4.8] | -10.8 [-16.9 to -4.4] | -5.0 [-11.6 to 2.1] | -12.4 [-18.3 to -6.1] | 9.2 [1.8 to 17.1]

ADVERSE EVENTS:
Time Frame: Adverse events are reported by treatment phase: Romosozumab treatment phase (Baseline [BL] to month 12 and 24); Denosumab extension phase (months 24 to 36); Romosozumab retreatment phase (months 36 to 48); Follow-on phase (months 48 to 72).
Description: The safety subset is based on actual treatment received. One participant randomized to placebo received 1 dose of romosozumab 70 mg in error was subsequently randomized to denosumab and then received romosozumab in the retreatment phase. Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed a 5% threshold
Groups:
- BL-Month 12: Placebo QM: Participants received placebo matching to romosozumab once a month (QM) administered subcutaneously for 12 months.
- BL-Month 12: Placebo Q3M: Participants received placebo matching to romosozumab once every 3 months (Q3M) administered subcutaneously for 12 months.
- BL-Month 12: Alendronate: Participants received open-label alendronate (ALN) 70 mg orally (PO) every week (QW) for 12 months.
- BL-Month12: Teriparatide: Participants received open-label teriparatide 20 μg subcutaneously every day (QD) for 12 months.
- BL-Month 12: Romosozumab 70 mg QM: Participants received double-blind romosozumab 70 mg subcutaneously every month for 12 months.
- BL-Month 12: Romosozumab 140 mg Q3M: Participants received double-blind romosozumab 140 mg subcutaneously once every 3 months for 12 months.
- BL-Month 12: Romosozumab 140 mg QM: Participants received double-blind romosozumab 140 mg subcutaneously every month for 12 months.
- BL-Month 12: Romosozumab 210 mg Q3M: Participants received double-blind romosozumab 210 mg Q3M subcutaneously for 12 months.
- BL-Month 12: Romosozumab 210 mg QM: Participants received double-blind romosozumab 210 mg QM subcutaneously for 12 months.
- BL-Month 24: Placebo QM: Participants received placebo matching to romosozumab QM administered subcutaneously for 24 months.
- BL-Month 24: Placebo Q3M: Participants received placebo matching to romosozumab Q3M administered subcutaneously for 24 months.
- BL-Month 24: ALN/Romosozumab 140 mg QM: Participants received open-label alendronate (ALN) 70 mg PO QW for 12 months. At month 12 participants transitioned to receive romosozumab 140 mg subcutaneously every month for an additional 12 months (months 12 to 24).
- BL-Month 24: Romosozumab 70 mg QM: Participants received double-blind romosozumab 70 mg subcutaneously every month for 24 months.
- BL-Month 24: Romosozumab 140 mg Q3M: Participants received double-blind romosozumab 140 mg subcutaneously once every 3 months for 24 months.
- BL-Month 24: Romosozumab 140 mg QM: Participants received double-blind romosozumab 140 mg subcutaneously every month for 24 months.
- BL-Month 24: Romosozumab 210 mg Q3M: Participants received double-blind romosozumab 210 mg Q3M subcutaneously for 24 months.
- BL-Month 24: Romosozumab 210 mg QM: Participants received double-blind romosozumab 210 mg QM subcutaneously for 24 months.
- Month 24-36: Placebo/Placebo: Participants who received placebo in the 24-month romosozumab treatment phase then received placebo to denosumab subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 24-36: ALN/Romosozumab/Placebo: Participants who received alendronate for the first 12 months and romosozumab 140 mg subcutaneously every month from months 12 to 24 received placebo to denosumab subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 24-36: ALN/Romosozumab/Denosumab: Participants who received alendronate for the first 12 months, romosozumab 140 mg subcutaneously every month from months 12-24 received denosumab 60 mg subcutaneously once every 6 months for 12 months during the denosumab extension phase.
- Month 36-48: Placebo/Placebo/Romosozumab: Participants who received placebo in the first 24-month romosozumab treatment phase and placebo to denosumab during months 24 to 36 then received romosozumab 210 mg subcutaneously QM in the 12-month romosozumab retreatment phase (months 36 to 48).
- Month 36-48: Placebo/Denosumab/Romosozumab: Participants who received placebo in the first 24-month romosozumab treatment phase and denosumab 60 mg during months 24 to 36 then received romosozumab 210 mg subcutaneously QM in the 12-month romosozumab retreatment phase (months 36 to 48).
- Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention: Participants who received romosozumab at any dose during the first 24 month treatment phase, denosumab 60 mg during months 24 to 36 and romosozumab 210 mg QM in months 36 to 48 then received no intervention during the 24-month follow-on phase (months 48-72).
- Month 48-72: Romosozumab/Placebo/Romosozumab/No: Participants who received romosozumab at any dose during the first 24 month treatment phase, placebo to denosumab during months 24 to 36 and romosozumab 210 mg QM in months 36 to 48 were assigned to the zoledronic acid treatment group, but received no intervention during the 24-month follow-on phase (months 48 to 72).
- Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic: Participants who received placebo in the 24-month romosozumab treatment phase, denosumab 60 mg Q6M from months 24 to 36 and romosozumab 210 mg QM from months 36 to 48 then received a single dose of open-label zoledronic acid 5 mg intravenously at month 48.
Arm/Group | BL-Month 12: Placebo QM | BL-Month 12: Placebo Q3M | BL-Month 12: Alendronate | BL-Month12: Teriparatide | BL-Month 12: Romosozumab 70 mg QM | BL-Month 12: Romosozumab 140 mg Q3M | BL-Month 12: Romosozumab 140 mg QM | BL-Month 12: Romosozumab 210 mg Q3M | BL-Month 12: Romosozumab 210 mg QM | BL-Month 24: Placebo QM | BL-Month 24: Placebo Q3M | BL-Month 24: ALN/Romosozumab 140 mg QM | BL-Month 24: Romosozumab 70 mg QM | BL-Month 24: Romosozumab 140 mg Q3M | BL-Month 24: Romosozumab 140 mg QM | BL-Month 24: Romosozumab 210 mg Q3M | BL-Month 24: Romosozumab 210 mg QM | Month 24-36: Placebo/Placebo | Month 24-36: Placebo/Denosumab | Month 24-36: ALN/Romosozumab/Placebo | Month 24-36: ALN/Romosozumab/Denosumab | Month 24-36: Romosozumab/Placebo | Month 24-36: Romosozumab/Denosumab | Month 36-48: Placebo/Placebo/Romosozumab | Month 36-48: Placebo/Denosumab/Romosozumab | Month 36-48: Romosozumab/Placebo/Romosozumab | Month 36-48: Romosozumab/Denosumab/Romosozumab | Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention | Month 48-72: Romosozumab/Placebo/Romosozumab/No | Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic | Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid | Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 3/30 | 4/20 | 4/51 | 5/54 | 5/50 | 3/52 | 2/49 | 3/53 | 6/51 | 5/30 | 4/20 | 8/51 | 9/50 | 8/52 | 8/49 | 6/53 | 7/51 | 2/18 | 1/17 | 2/19 | 0/19 | 3/90 | 8/89 | 0/12 | 1/15 | 4/72 | 3/68 | 8/51 | 0/3 | 1/11 | 1/12 | 9/56 | 1/8
Other Adverse Events (participants affected / at risk) | 25/30 | 19/20 | 38/51 | 36/54 | 46/50 | 40/52 | 41/49 | 45/53 | 40/51 | 28/30 | 20/20 | 49/51 | 48/50 | 47/52 | 46/49 | 51/53 | 47/51 | 15/18 | 15/17 | 12/19 | 15/19 | 57/90 | 59/89 | 12/12 | 11/15 | 53/72 | 55/68 | 34/51 | 1/3 | 10/11 | 8/12 | 44/56 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BL-Month 12: Placebo QM (N=30) | BL-Month 12: Placebo Q3M (N=20) | BL-Month 12: Alendronate (N=51) | BL-Month12: Teriparatide (N=54) | BL-Month 12: Romosozumab 70 mg QM (N=50) | BL-Month 12: Romosozumab 140 mg Q3M (N=52) | BL-Month 12: Romosozumab 140 mg QM (N=49) | BL-Month 12: Romosozumab 210 mg Q3M (N=53) | BL-Month 12: Romosozumab 210 mg QM (N=51) | BL-Month 24: Placebo QM (N=30) | BL-Month 24: Placebo Q3M (N=20) | BL-Month 24: ALN/Romosozumab 140 mg QM (N=51) | BL-Month 24: Romosozumab 70 mg QM (N=50) | BL-Month 24: Romosozumab 140 mg Q3M (N=52) | BL-Month 24: Romosozumab 140 mg QM (N=49) | BL-Month 24: Romosozumab 210 mg Q3M (N=53) | BL-Month 24: Romosozumab 210 mg QM (N=51) | Month 24-36: Placebo/Placebo (N=18) | Month 24-36: Placebo/Denosumab (N=17) | Month 24-36: ALN/Romosozumab/Placebo (N=19) | Month 24-36: ALN/Romosozumab/Denosumab (N=19) | Month 24-36: Romosozumab/Placebo (N=90) | Month 24-36: Romosozumab/Denosumab (N=89) | Month 36-48: Placebo/Placebo/Romosozumab (N=12) | Month 36-48: Placebo/Denosumab/Romosozumab (N=15) | Month 36-48: Romosozumab/Placebo/Romosozumab (N=72) | Month 36-48: Romosozumab/Denosumab/Romosozumab (N=68) | Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention (N=51) | Month 48-72: Romosozumab/Placebo/Romosozumab/No (N=3) | Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid (N=11) | Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic (N=12) | Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid (N=56) | Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid (N=8)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mycobacterium kansasii infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hysterocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BL-Month 12: Placebo QM (N=30) | BL-Month 12: Placebo Q3M (N=20) | BL-Month 12: Alendronate (N=51) | BL-Month12: Teriparatide (N=54) | BL-Month 12: Romosozumab 70 mg QM (N=50) | BL-Month 12: Romosozumab 140 mg Q3M (N=52) | BL-Month 12: Romosozumab 140 mg QM (N=49) | BL-Month 12: Romosozumab 210 mg Q3M (N=53) | BL-Month 12: Romosozumab 210 mg QM (N=51) | BL-Month 24: Placebo QM (N=30) | BL-Month 24: Placebo Q3M (N=20) | BL-Month 24: ALN/Romosozumab 140 mg QM (N=51) | BL-Month 24: Romosozumab 70 mg QM (N=50) | BL-Month 24: Romosozumab 140 mg Q3M (N=52) | BL-Month 24: Romosozumab 140 mg QM (N=49) | BL-Month 24: Romosozumab 210 mg Q3M (N=53) | BL-Month 24: Romosozumab 210 mg QM (N=51) | Month 24-36: Placebo/Placebo (N=18) | Month 24-36: Placebo/Denosumab (N=17) | Month 24-36: ALN/Romosozumab/Placebo (N=19) | Month 24-36: ALN/Romosozumab/Denosumab (N=19) | Month 24-36: Romosozumab/Placebo (N=90) | Month 24-36: Romosozumab/Denosumab (N=89) | Month 36-48: Placebo/Placebo/Romosozumab (N=12) | Month 36-48: Placebo/Denosumab/Romosozumab (N=15) | Month 36-48: Romosozumab/Placebo/Romosozumab (N=72) | Month 36-48: Romosozumab/Denosumab/Romosozumab (N=68) | Month 48-72: Romosozumab/Denosumab/Romosozumab/No Intervention (N=51) | Month 48-72: Romosozumab/Placebo/Romosozumab/No (N=3) | Month 48-72: Placebo/Placebo/Romosozumab/Zoledronic Acid (N=11) | Month 48-72: Placebo/Denosumab/Romosozumab/Zoledronic (N=12) | Month 48-72: Romosozumab/Placebo/Romosozumab/Zoledronic Acid (N=56) | Month 48-72: Romosozumab/Denosumab/Romosozumab/Zoledronic Acid (N=8)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presbyacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 3 | 2 | 3 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 5 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 4 | 2 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 4 | 0 | 1 | 1 | 1 | 1 | 1 | 4 | 4 | 0 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 3 | 2 | 5 | 2 | 5 | 5 | 2 | 3 | 0 | 4 | 6 | 3 | 5 | 5 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 3 | 2 | 4 | 0 | 0 | 3 | 2 | 3 | 5 | 3 | 4 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 5 | 1 | 0 | 0 | 0 | 3 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 4 | 0 | 1 | 3 | 0 | 2 | 1 | 3 | 6 | 0 | 1 | 5 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 5 | 9 | 1 | 3 | 0 | 0 | 3 | 0 | 0 | 9 | 1 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 3 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 5 | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 6 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 4 | 1 | 5 | 1 | 2 | 1 | 1 | 6 | 6 | 1 | 7 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 9 | 0
Injection site bruising (General disorders) | 2 | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 4 | 3 | 0 | 0 | 2 | 4 | 3 | 5 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 3 | 3 | 0 | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Borrelia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 2 | 5 | 5 | 3 | 1 | 2 | 2 | 2 | 6 | 6 | 5 | 5 | 3 | 4 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 3 | 0 | 1 | 2 | 3 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 1 | 3 | 6 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 2 | 5 | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema migrans (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2 | 1 | 3 | 2 | 4 | 5 | 8 | 2 | 1 | 4 | 4 | 2 | 4 | 5 | 9 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 3 | 3 | 2 | 1 | 1 | 2 | 4 | 5 | 3 | 10 | 7 | 3 | 4 | 5 | 8 | 0 | 1 | 0 | 1 | 2 | 4 | 3 | 1 | 8 | 7 | 1 | 0 | 0 | 2 | 8 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 3 | 4 | 19 | 10 | 13 | 5 | 9 | 8 | 4 | 10 | 20 | 14 | 17 | 10 | 14 | 1 | 1 | 3 | 4 | 7 | 10 | 3 | 3 | 8 | 11 | 4 | 0 | 2 | 2 | 4 | 2
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 4 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 3 | 3 | 2 | 0 | 2 | 0 | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 0 | 3 | 0 | 2 | 2 | 2 | 1 | 2 | 3 | 7 | 2 | 4 | 6 | 7 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 1 | 4 | 1 | 1 | 0 | 6 | 2 | 0 | 3 | 7 | 3 | 3 | 2 | 8 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 4 | 3 | 0 | 3 | 3 | 5 | 5 | 3 | 0 | 7 | 5 | 4 | 4 | 9 | 6 | 0 | 1 | 1 | 0 | 5 | 1 | 0 | 0 | 4 | 1 | 6 | 0 | 0 | 0 | 1 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 0 | 2 | 1 | 3 | 5 | 1 | 1 | 0 | 4 | 0 | 2 | 4 | 5 | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 1 | 2 | 3 | 2 | 1 | 1 | 2 | 0 | 7 | 4 | 3 | 7 | 3 | 4 | 1 | 0 | 1 | 1 | 3 | 4 | 0 | 1 | 3 | 4 | 0 | 1 | 0 | 0 | 4 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 2 | 2 | 0 | 2 | 4 | 6 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 4 | 0 | 0 | 1 | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2 | 2 | 1 | 1 | 0 | 2 | 2 | 1 | 3 | 3 | 1 | 3 | 1 | 4 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 5 | 8 | 7 | 6 | 5 | 2 | 8 | 3 | 11 | 10 | 8 | 6 | 9 | 6 | 1 | 0 | 1 | 3 | 2 | 6 | 2 | 0 | 6 | 11 | 1 | 1 | 1 | 0 | 8 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 6 | 3 | 4 | 4 | 7 | 7 | 3 | 7 | 2 | 12 | 8 | 8 | 12 | 9 | 5 | 1 | 1 | 1 | 2 | 1 | 4 | 2 | 0 | 6 | 8 | 2 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 8 | 0 | 2 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2 | 4 | 2 | 2 | 3 | 1 | 3 | 0 | 3 | 8 | 3 | 2 | 4 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 4 | 2 | 3 | 3 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 2 | 4 | 0 | 1 | 0 | 3 | 7 | 2
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 3 | 2 | 2 | 2 | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 5 | 1 | 5 | 2 | 6 | 3 | 5 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 2 | 1 | 3 | 0 | 1 | 0 | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 5 | 10 | 7 | 5 | 3 | 6 | 4 | 0 | 3 | 12 | 8 | 6 | 5 | 6 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 4 | 2 | 1 | 0 | 1 | 1 | 4 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Thoracic spine flattening (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 5 | 3 | 3 | 1 | 1 | 2 | 3 | 2 | 4 | 4 | 6 | 1 | 2 | 4 | 2 | 3 | 0 | 1 | 1 | 2 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Facial neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 3 | 3 | 3 | 7 | 3 | 3 | 5 | 5 | 3 | 6 | 5 | 8 | 3 | 4 | 7 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 3 | 5 | 3 | 1 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 2 | 0 | 0 | 1 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Breast calcifications (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 0 | 8 | 3 | 4 | 1 | 5 | 3 | 1 | 6 | 8 | 5 | 8 | 3 | 8 | 1 | 0 | 0 | 1 | 3 | 4 | 2 | 0 | 3 | 3 | 3 | 0 | 1 | 2 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 4 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 4 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intraocular lens implant (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Tooth repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 1 | 2 | 3 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 4 | 4 | 6 | 3 | 4 | 0 | 0 | 0 | 0 | 4 | 3 | 2 | 1 | 3 | 6 | 1 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.